CLINICAL TRIAL: NCT02961413
Title: A Multi-center, Prospective, Non-interventional Cohort Study on Drug Induced Liver Injury in Mainland China
Brief Title: A Prospective Cohort Study on Drug-induced Liver Injury in China（DILI-P）
Acronym: DILI-P
Status: Recruiting | Type: Observational
Sponsor: Drug Induced Liver Disease Study Group (Other)
Responsible Party: Sponsor
Other Study IDs: 2012ZX09303-002
Record Dates: First submitted 2016-10-24; First posted 2016-11-11 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Drug-induced Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, histology, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- cohort 1: Compound glycyrrhizin tablets / injection
- cohort 2: Isoglycyrrhizinate magnesium injection / diammonium glycyrrhizinate enteric-coated capsules
- cohort 3: Bicyclol
- cohort 4: Silibinin capsules
- cohort 5: Ursodeoxycholic acid capsules
- cohort 6: N- acetylcysteine

SUMMARY:
This is a multi-center, prospective, non-interventional cohort study .

Its primary objectives are:

1. assess DILI patients' clinical characteristics, disease progression and influencing factors in clinical practice;
2. learn about suspected drug caused DILI,rechallenging, liver biochemical abnormalities mode, etc.

DETAILED DESCRIPTION:
The main purpose of this study is to understand patients with DILI clinical outcome and influencing factors in China's second and tertiary general hospitals (including Western medicine hospital, Chinese medicine hospital andIntegrated traditional Chinese and Western Medicine Hospital) and vulnerabilities of drug-induced liver injury specialist hospital (tuberculosis hospital, Pulmonary, etc.) in mainland.

The main purpose

1. assess the DILI patients' clinical outcomes and influencing factors in the real world;
2. learn about suspected drug caused DILI,rechallenging, liver biochemical abnormalities mode, etc.

Secondary objectives

1. assess the compliance of the DILI practice to the 2015 vision of the DILI guidelines in china.;
2. evaluate the histological features of DILI patients;
3. assessment DILI characteristics, prognosis and influencing factors in specific populations(such as the elderly, children with underlying liver disease background, etc.)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DILI patients with various types and severity according to the 2015 version of the Chinese DILI treatment guidelines
* RUCAM ≥6, or RUCAM between 3-5 is required by the three experts determined that the drug-induced liver injury
* patient can provide informed consent form

Exclusion Criteria:

* non-drug-induced liver injury

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with drug-induced liver injury
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-04; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Disease progression of DILI (drug-induced liver injury ), i.e. death, liver failure, chronic DILI, recover | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Mao, Study Chair — RenJi Hospital; Chengwei Chen, Study Chair — No.85 Hospital of PLA; Xingfang Li, Principal Investigator — Pulmonary Hospital of Lanzhou; Yiling Li, Principal Investigator — First Hospital of China Medical University; Dongliang Li, Principal Investigator — Fuzhou General Hospital; Suocai Zhang, Principal Investigator — Changzhou Third People 's Hospital; Rongxia Sang, Principal Investigator — First Hospital of Shijiazhuang City; Zhihui Li, Principal Investigator — Hebei Chest Hospital; Feng Sun, Principal Investigator — First Affiliated Hospital of Heilongjiang Chinese Medicine University; Wushu Yan, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Yanqin Wu, Principal Investigator — Bazhou People 's Hospital; Xu Lian, Principal Investigator — Mudanjiang Red Flag Hospital; Mingfang Wang, Principal Investigator — Pingdingshan People's Hospital No.1; Yanrong Shi, Principal Investigator — General Hospital of Pingdingshan Coal Industry Company; Hongwei Chen, Principal Investigator — Luoyang Central Hospital; Ximei Wang, Principal Investigator — Third Hospital Affiliated to Henan University of Science and Technology; Hongling Liu, Principal Investigator — The First People's Hospital of Luoyang; Renping Li, Principal Investigator — The Second Hospital Affiliated to Henan University of Science and Technology; Zhengsheng Zou, Principal Investigator — Beijing 302 Hospital; Jiguang Ding, Principal Investigator — The Third Affiliated Hospital of Wenzhou Medical University; Yanjun Guo, Principal Investigator — Daqing oilfield general hospital; Weixin He, Principal Investigator — The No.123 Hospital of Chinese People's Liberation Army; Wufang Qi, Principal Investigator — Tianjin First Central Hospital; Yuqin Xu, Principal Investigator — The No.211 Hospital of Chinese People's Liberation Army; Jing Zhang, Principal Investigator — Beijin Youan Hospital,Capital Medical University; Peilan Zong, Principal Investigator — Jiangxi Chest Hospital; Yuefei Shen, Principal Investigator — The First People's Hospital of Hangzhou Xiaoshan District; Chunyan Zhou, Principal Investigator — Infectious Diseases Hospital of Shangqiu; Baijing Ding, Principal Investigator — The Second People's Hospital of Wuhu; Liyun Chen, Principal Investigator — Wuhu Third People's Hospital; Yongze Guo, Principal Investigator — Affiliated Hospital of Hebei University of Engineering; Haibin Wang, Principal Investigator — Fifth Hospital of Shijiazhuang City; Hui Guo, Principal Investigator — First Teaching Hospital of Tianjin University of Traditional Chinese Medicine; Hongling Liu, Principal Investigator — Beijing 302 Hospital; Yingjian Zhang, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Qing Mao, Principal Investigator — Southwest Hospital, China; Liaoyun Zhang, Principal Investigator — The First Affiliated Hospital of Shanxi Medical University; Jiawei Gen, Principal Investigator — First People's Hospital of Yunnan Province; Weize Zuo, Principal Investigator — The First Affiliated Hospital of Medical College,Shihezi University; Xia Zhang, Principal Investigator — Nanjing Chest Hospital; Xuan Zhu, Principal Investigator — The First Affiliated Hospital of Nanchang University; Feng Shuai, Principal Investigator — Linyi People's Hospital; Kunyun Yang, Principal Investigator — Hunan Chest Hospital; Chuanwu Zhu, Principal Investigator — The Fifth People,Hospital of Suzhou; Wei Ge, Principal Investigator — Renmin Hospital of Wuhan University; Xiaojin Wang, Principal Investigator — 85 Hospital of People's Liberation Army; Jiajun Liu, Principal Investigator — The First Affiliated Hospital of Xiamen University; Yan Huang, Principal Investigator — Xiangya Hospital of Central South University; Fangping He, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Xinmin Zhou, Principal Investigator — Xijing Hospital; Aiqing Lin, Principal Investigator — The First Affiliated Hospital of Inner Mongolia University of Science and Technology; Xiaojing Jiang, Principal Investigator — Wuhan General Hospital of Guangzhou Military; Qing Xie, Principal Investigator — Ruijin Hospital; Qingge Zhang, Principal Investigator — Xingtai People's Hospital; Yanyan Yu, Principal Investigator — Peking University First Hospital; Jing Yuan, Principal Investigator — Shenzhen Third People's Hospital; Shiwu Ma, Principal Investigator — Kunming General Hospital of Chengdu Military Area Command; Jun Chen, Principal Investigator — Second Xiangya Hospital of Central South University; Qinghua Yao, Principal Investigator — Zhejiang Cancer Hospital; Yihong Zhang, Principal Investigator — The No.457 Hospital of Chinese People's Liberation Army; Qi Wang, Principal Investigator — Second Hospital of Shanxi Medical University; Xiaozhong Wang, Principal Investigator — Xinjiang Autonomous Region Hospital of TCM; Yongwen Ma, Principal Investigator — Daqing Longnan Hopital; Fangfang Lv, Principal Investigator — Sir Run Run Shaw Hospital; Xiaojun Zhang, Principal Investigator — Ankang City Central Hospital; Riwang Hu, Principal Investigator — The Fouth People's Hospital of Datong; Yi Song, Principal Investigator — Chongqing Traditional Chinese Medicine Hospital; Peng Hu, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Wen Xie, Principal Investigator — Beijing Ditan Hospital; Yongguo Li, Principal Investigator — First Affiliated Hospital of Harbin Medical University; Haiyan Jin, Principal Investigator — Yanbian University Hospital; Zheng Li, Principal Investigator — The First People's Hospital of Qinzhou; Shuixiang He, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Lei Li, Principal Investigator — Anhui Provincial Hospital; Junqi Niu, Principal Investigator — The First Affiliated Hospital of Jilin University; Bin Jiang, Principal Investigator — The Second People's Hospital of Liaoyuan; Jing You, Principal Investigator — First Affiliated Hospital of Kunming Medical University; Youqin Yan, Principal Investigator — WUHAN NO.7 HOSPITAL; Lvye Xv, Principal Investigator — General Hospital of The Yangtze River Shipping; Changyong Zhang, Principal Investigator — Wuhan Mental Health Centre; Guanghua Xv, Principal Investigator — Ya'nan University Affiliated Hospital; Hongbin Li, Principal Investigator — The First Affiliated Hospital of Anhui Medical University; Yongfeng Yang, Principal Investigator — The Second Hospital of Nanjing Medical University; Xilian Dong, Principal Investigator — Yuncheng Central Hospital; Xuefeng Su, Principal Investigator — LinFen People's Hospital; Mudan Yang, Principal Investigator — Shanxi Provincial Cancer Hospital; Zhen Ma, Principal Investigator — The Affiliated Hospital of Inner Mongolia Medical University; Hong Tang, Principal Investigator — West China Hospital; Chenghai Liu, Principal Investigator — Shanghai Shuguang Hospital; Zhenyu Yan, Principal Investigator — South China University of Science And Technology Affiliated Hospital; Fei Qiao, Principal Investigator — Jiangsu province hospital of TCM; Xingxiang Yang, Principal Investigator — Sichuan Province Hospital; Jinjun Chen, Principal Investigator — Nanfang Hospital, Southern Medical University; Weihong Sha, Principal Investigator — Guangdong Provincial People's Hospital; Jie Jin, Principal Investigator — First People's Hospital of Hangzhou; Feng Lin, Principal Investigator — Hainan General Hospital; Guoqi Zheng, Principal Investigator — Cangzhou Central Hospital; Jiyao Wang, Principal Investigator — Zhong Shan Hospital; Lin Chen, Principal Investigator — LanZhou University; Dongliang Yang, Principal Investigator — Tongji Medical College of Huazhong University of Science and Technology; Li Chen, Principal Investigator — The Center Hospital Of Maanshan; Guizhou Zou, Principal Investigator — The Second Hospital of Anhui Medical University; Yong Wang, Principal Investigator — Fuyang First People's Hospital; Lianqing Lou, Principal Investigator — Yiwu Central Hospital; Huaming Li, Principal Investigator — The Third People's Hospital of Hangzhou; Shifang Chen, Principal Investigator — Huzhou Central Hospital; Zhifen Pan, Principal Investigator — Affiliated Hospital of Jiaxing University; Wenlong Zheng, Principal Investigator — Hangzhou Hospital of Traditional Chinese Medicine; Jingbo Pei, Principal Investigator — Hangzhou Xiaoshan Hospital of Traditional Chinese Medicine; Feng Guo, Principal Investigator — Hangzhou Xiaoshan First People's Hospital; Feng Qian, Principal Investigator — Dongyang People's Hospital; Jianzheng Mao, Principal Investigator — Zhejiang Quhua Hospital; Ahuo Ma, Principal Investigator — Shaoxing People's Hospital; Qinhong Zheng, Principal Investigator — People's Hospital of Quzhou; Jufen Xu, Principal Investigator — Tongxiang First People's Hospital; Jiemin Hong, Principal Investigator — Ningbo Yinzhou No.2 Hospital; Jianwei Shen, Principal Investigator — Ningbo Medical Center Lihuili Eastern Hospital; Yunsong Qian, Principal Investigator — Ningbo No.2 Hospital; Weihong Du, Principal Investigator — Jinhua Central Hospital; Jiaxin Liu, Principal Investigator — Huzhou Hospital of Traditional Chinese Medicine; Qingjing Ru, Principal Investigator — Zhejiang Construction Hospital; Chunsheng Zhao, Principal Investigator — The No.98 Hospital of Chinese People's Liberation Army; Yinxia Hao, Principal Investigator — Baoding First Central Hospital; Li Sun, Principal Investigator — Xi'an No.3 Hospital; Wenlei Hu, Principal Investigator — Le Qin People's Hospital; Shuangsuo Dang, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University; Yu Chen, Principal Investigator — Zhengzhou No.6 People's Hospital; Zhaoxia Liu, Principal Investigator — First Affiliated Hospital of Heilongjiang Chinese Medicine University; Yang Pan, Principal Investigator — Heilongjiang Provincial Hospital of Traditional Chinese Medicine; Yi Shen, Principal Investigator — Dandong City Infectious Disease Hospital; Xia Li, Principal Investigator — Baoding City Infectious Disease Hospital; Qian Zhong, Principal Investigator — Anshan Central Hospita; Zhixiong Fang, Principal Investigator — Xiangtan Central Hospita; Xiaoping Xu, Principal Investigator — Xiangxi Autonomous Prefecture People's Hospital; Sihai Li, Principal Investigator — The First People's Hospital of YueYang; Hui Tian, Principal Investigator — The People's Hospital of Xuancheng City; Shiquan Ka, Principal Investigator — The First People's Hospital of Lanzhou City; Dongfang Li, Principal Investigator — Anhui Province Chest Hospital; Yuqiang Nie, Principal Investigator — Guangzhou First People's Hospital; Yan Song, Principal Investigator — Heilongjiang Mudanjiang Nanshan Hospital; Xiaoyan Guo, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University; Caiyan Zhao, Principal Investigator — Hebei Medical University Third Hospital; Yuemin Nan, Principal Investigator — Hebei Medical University Third Hospital; Dingguo Wang, Principal Investigator — People 's Hospital of Kaizhou District, Chongqing City; Li Wang, Principal Investigator — Public Health Clinical Center of Chengdu; Lixin Tong, Principal Investigator — First Hospital of Hebei Medical University; Hao Wu, Principal Investigator — West China Hospital,Huaxi University; Shurui Piao, Principal Investigator — Jinshan Hospital Fudan University; Lvfeng Yao, Principal Investigator — Meng Chao Liver and Gallbladder Hospital of Fujian Medical University; Yanqing Tian, Principal Investigator — Affiliated Hospital of Hebei University; Zhenbin Hu, Principal Investigator — The First Affiliated Hospital of Guangxi University of Chinese Medicine; Caisheng Wang, Principal Investigator — No.2 Hospital Of Huhhot; Xiaoyan Wang, Principal Investigator — The Third Xiangya Hospital of Central South University; Feng Jin, Principal Investigator — Shandong Provincial Chest Hospital; Yanbo Jiang, Principal Investigator — Donggang Center Hospital; Zhiqiang Wang, Principal Investigator — The 3Th People's Hospital Of Hengshui; Yu Xiong, Principal Investigator — Shandong Provincial Chest Hospital; Xinmei Guo, Principal Investigator — Shandong Provincial Chest Hospital; Yan Zhuang, Principal Investigator — People's Hospital Of Nongan county; Chaoren Zhao, Principal Investigator — Shandong Provincial Chest Hospital; Zhonghua Zhao, Principal Investigator — Tuberculosis Department, Shandong Provincialchest Hospital; Meiying Lin, Principal Investigator — Tuberculosis Department, Shandong Provincialchest Hospital; Jihong Yang, Principal Investigator — Affiliated Hospital of Hebei University; Jingyi Zhang, Principal Investigator — The Center Hospital Of Maanshan; Sangen Chen, Principal Investigator — People's Hospital Of Jinxian county; Yongping Pan, Principal Investigator — The Fourth Affiliated Hospital of Nanchang University; Ruipu Li, Principal Investigator — Second Central Hospital of Baoding; Xueshan Tao, Principal Investigator — Lushan Tuberculosis Prevention and Control Hospital; Shilin Qu, Principal Investigator — Ganzhou People's Hospital; Jie Liu, Principal Investigator — Jingzhou Chest Hospital; Diefeng Yin, Principal Investigator — People's Hospital Of Luxi county; Jianfeng Wu, Principal Investigator — Chinese Medicine Hospital of Gao'an City; Xueqiang Jiang, Principal Investigator — Sinopharm Dongfeng General Hospital; Jianwei Yang, Principal Investigator — Fujian Cancer Hospital; Yong Yang, Principal Investigator — The 94th Hospital of the People's Liberation Army; Chengyun Yang, Principal Investigator — People's Hospital Of Nanchang county; Shengjun Li, Principal Investigator — People's Hospital Of Xunyang; Jizhu Zhang, Principal Investigator — The Third People's Hospital Of Weifang; Jianjun Zhao, Principal Investigator — The Third People's Hospital Of Weifang; Gang Wu, Principal Investigator — The Third People's Hospital Of Jiujiang City; Yong Li, Principal Investigator — Fengyang County People's Hospital; Yansheng Sun, Principal Investigator — Infectious Disease Hospital Of Heilongjiang Province; Xiong Tang, Principal Investigator — Third People's Hospital Of Jiujiang City; Shousong Zhao, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University; Jiandao Zhang, Principal Investigator — Lingbi County People's Hospital; Long Yu, Principal Investigator — Liu'an People's Hospital; Weihua Xun, Principal Investigator — Shexian People's Hospital; Yong Jia, Principal Investigator — Anhui Provincial Hospital; Yi Li, Principal Investigator — Anhui Provincial Hospital Infectious Hospital; Zhengmao Yang, Principal Investigator — The Second People's Hospital Of Lanzhou City; Jianmin Liu, Principal Investigator — Zhuzhou No.2 Hospital; Huafa Yin, Principal Investigator — The First Affiliated Hospital of Anhui Medical University; Meilong Ding, Principal Investigator — Anhui Province Xuancheng City Central Hospital; Shanlou Hu, Principal Investigator — People's Hospital Of Dongzhi county; Yi Ding, Principal Investigator — Xiaoxian People's Hospital; Weidong Fang, Principal Investigator — Huangshan City People's Hospital; Liu Hong, Principal Investigator — Anhui Wuhu County Hospital; Xiaorong Xu, Principal Investigator — Bozhou Hospital of Traditional Chinese Medicine; Delian Wu, Principal Investigator — Suzhou Hospital Affiliated To Anhui Medical University; Yong Huang, Principal Investigator — The Second People's Hospital of Hefei; Qiliang Tan, Principal Investigator — Dazhou Central Hospital; Songqing Liao, Principal Investigator — Huainanchaoyang Hospital; Bin Yao, Principal Investigator — The People's Hospital Huaibei; Shuiqing Jiang, Principal Investigator — Huainan First People's Hospital; Yanmin Wang, Principal Investigator — Infectious Disease Hospital Of Baishan; Lei Zhang, Principal Investigator — Anhui Chest Hospital; Wenhong Lin, Principal Investigator — Anhui Chest Hospital; Wengang Zhang, Principal Investigator — Tonghua Central Hospital; Chongfeng Gu, Principal Investigator — The Ninth People's Hospital Of Jilin; Zhe Zhang, Principal Investigator — Jilin Tuberculosis Prevention and Control Institute; Junfeng Wang, Principal Investigator — Jixijikuang Hospital; Jie Zhou, Principal Investigator — Tianjin Tuberculosis Prevention and Control Center; Guomin Tang, Principal Investigator — Renmin Hospital Of Shayang; Zhuo Li, Principal Investigator — Baiyupao Hospital; Guohui Zhu, Principal Investigator — The Third People's Hospital Of Weifang; Xingping Liu, Principal Investigator — The Third People's Hospital Of Weifang; Jingen Wang, Principal Investigator — Zhangshu People's Hospital; Xinyan Zhao, Principal Investigator — Beijing Friendship Hospital; Hongliang Liang, Principal Investigator — Avic 363 Hospital; Lijun Liu, Principal Investigator — Yiyang Central Hospital; Fangchun Li, Principal Investigator — Fengcheng People's Hospital; Jianwei Zhou, Principal Investigator — Xiangdong Hospital Hunan Normal University; Zhongrui Su, Principal Investigator — Zhangjiajie City People's Hospital; Wei Xiao, Principal Investigator — The Third Xiangya Hospital of Central South University; Bohui Yuan, Principal Investigator — Qitaihe Coal Mine Hospital; Chun Yang, Principal Investigator — Beilun People's Hospital; Gaizhi Zhang, Principal Investigator — Luohe Psychiatric Hospital; Ming Li, Principal Investigator — No.2 People's Hospital of Fuyang City; Zhixue Zhang, Principal Investigator — Qiqihar Tuberculosis Prevention and Control Center; Wei Yue, Principal Investigator — The First People's Hospital of Yunnan; Li Zhou, Principal Investigator — Ningbo Medical Center Lihuili Eastern Hospital; Xiaoqing Li, Principal Investigator — Anqing Municipal Hospitalis; Chunge Tian, Principal Investigator — Dengzhou Central Hospital; Tianming Wang, Principal Investigator — No.1 People's Hospital Of Zhumadian; Ji'ao Han, Principal Investigator — People's Hospital of Zhengzhou University; Jingxia Ma, Principal Investigator — People's Hospital Of Xinye; Jie Bao, Principal Investigator — The First People's Hospital of Xinmi; Jianhui Sun, Principal Investigator — Weihui People's Hospital; Xiaoju Luo, Principal Investigator — Yuanyang Central Hospital; Weili Niu, Principal Investigator — The Third People's Hospital Of Hebi; Ming Wang, Principal Investigator — Hepatobiliary Hospital Of Jilin; Yiwen Qiao, Principal Investigator — Dengzhou Hospital of TCM; Chuan Zhao, Principal Investigator — Suining Infectious Diseases Hospital; Xiaoqian Zhang, Principal Investigator — Anhui Mental Health Center; Jingchao Guo, Principal Investigator — Wugang People's Hospital; Weihua Liu, Principal Investigator — General Hospital of Heilongjiang Provincial Agricultural Reclamation Bureau; Feng Wu, Principal Investigator — Baoji People's Hospital; Man Chen, Principal Investigator — Taian Enliang Hospital; Hong Wu, Principal Investigator — Xiuyan Central Hospital; Shansong Bai, Principal Investigator — Anshan Mental Health Center; Xiuying Men, Principal Investigator — General Hospital Of Liaohe Oilfield; Yanhua Jiang, Principal Investigator — Tiefa Coal Group General Hospital; Junzu Yang, Principal Investigator — The People's Hospital Of Lingchengqu; Haiyan Zhou, Principal Investigator — Baoshan Hospital Of Chifeng; Yu Feng, Principal Investigator — The Third Affiliated Hospital of Jinzhou Medical University; Yihua Song, Principal Investigator — Liaoyang City Central Hospital; Tao Yang, Principal Investigator — Panshan Mental Rehabilitation Hospital; Yueping Li, Principal Investigator — Wafangdian Central hospital; Guosheng Jiang, Principal Investigator — People's Hospital Of Ningjinxian; Bo Zhang, Principal Investigator — Taian City Central Hospital; Shujun Geng, Principal Investigator — Hebei Chest Hospital; Jin Huang, Principal Investigator — The Second People's Hospital Of Changzhou; Fengming Yin, Principal Investigator — The 169th Hospital Of P.L.A.; Weiguo He, Principal Investigator — Public Health Affiliated Hospital,University Of South China; Zhefeng Zhong, Principal Investigator — Affiliated Nanhua Hospital，University Of South China; Yuan Yang, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Guoping Fang, Principal Investigator — The Third People's Hospital Of Changzhou; Qiang Miao, Principal Investigator — Tonghua Tuberculosis Prevention and Control Center; Xin'guang Huang, Principal Investigator — The Fourth People's Hospital of Chenzhou; Duanbao Tian, Principal Investigator — The Fourth People's Hospital Of Zibo; Yaoming Yuan, Principal Investigator — People's Hospital Of Shishou; Yuzi Lin, Principal Investigator — Yanji Tuberculosis Prevention and Control Center; Ligang Chen, Principal Investigator — Dunhua Tuberculosis Prevention and Control Center; Yu Zhang, Principal Investigator — Huichun Tuberculosis Prevention and Control Center; Chunrong Li, Principal Investigator — Yanji Brain Hospital; Aimin Wu, Principal Investigator — Yanji Brain Hospital; Xiangzhu Bai, Principal Investigator — Antu Tuberculosis Prevention and Control Center; Shaorong Deng, Principal Investigator — People's Hospital Of Zhongxiang; Shaoguang Yang, Principal Investigator — Tianjin Xiqing Hospital; Guohong Ge, Principal Investigator — People's Hospital Of Zhenjiang; Xuebing Yan, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Sheng Huang, Principal Investigator — People's Hospital Of Songzi; Gongying Chen, Principal Investigator — The Affiliated Hospital of Hangzhou Normal University; Ping Li, Principal Investigator — Tianjin Second People's Hospital; Jiehua Li, Principal Investigator — The First Affiliated Hospital of Anhui Medical University; Weiwei Kang, Principal Investigator — Beijing YouAn Hospital
Locations (1):
- Renji hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No